CLINICAL TRIAL: NCT04250610
Title: Postoperative Delirium in Poland - a Survey Assessing the Level of Knowledge of the POD Problem Among the Staff of Anaesthesiology and Intensive Care Departments.
Brief Title: Survey Assessing the Level of Knowledge of Postoperative Delirium in Poland.
Acronym: PODinPOL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Katarzyna Kotfis, Principal Investigator, Pomeranian Medical University Szczecin
Other Study IDs: KB-0012/06/01/2020/Z
Record Dates: First submitted 2020-01-30; First posted 2020-01-31 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Postoperative Delirium
Keywords: Postoperative delirium; POD; Anesthetics; Neurocognitive Disorders; Central Nervous System; Confusion; Neurologic Manifestations
MeSH Terms: conditions — Emergence Delirium; Neurocognitive Disorders; Confusion; Neurologic Manifestations | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — On-line survey.

SUMMARY:
Postoperative Delirium (POD) is one of the most common complications occurring after surgery with an incidence ranging from 4 to 53%. It may lead to increased postoperative morbidity and mortality, with loss of independence and cognitive dysfunction in certain groups of patients. Aiming to reduce the incidence of POD and improve the outcome of patients diagnosed with POD, it is necessary to raise awareness regarding POD. The most important issue are: identification of risk factors, improved monitoring, necessary prevention and adequate treatment. The Polish Society of Anaesthesiology and Intensive Therapy (PTAiIT) has made an attempt to improve the situation in Poland by testing the implementation of official POD guidelines published by the European Society of Anesthesiology in year 2017. While the guidelines provide recommendations for daily practice it is necessary to identify the degree of their implementation in each country. Therefore survey has been prepared regarding postoperative delirium in Poland. This Survey has been submitted to the Bioethical Committee of the Pomeranian Medical University in Szczecin (Poland) and received a waiver due to the non-interventional, observational character of the study (decision no. KB-0012/06/01/2020/Z).

ELIGIBILITY:
Inclusion Criteria:

* Specialists and residents working in the field of anesthesiology and intensive therapy, anesthesiology nurses who respond to an invitation to an on-line survey of the Polish Society of Anesthesiology and Intensive Therapy (PTAiIT)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Specialists and residents working in the field of anesthesiology and intensive therapy, members of the Polish Society of Anesthesiology and Intensive Therapy (PTAiIT).
Sampling Method: Probability Sample
Enrollment: 460 (Estimated)
Dates: Start 2020-02-27 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Status of diagnosis of postoperative delirium | Up to 2 months
  Answers of PTAiIT-members regarding instruments used to diagnose postoperative delirium. Anonymous on-line survey including Multiple Choice Questions, Closed and Open Questions.

SECONDARY OUTCOMES:
Identification of postoperative delirium risk factors | Up to 2 months
  Answers of PTAiIT-members regarding risk factors of postoperative delirium. Anonymous on-line survey including Multiple Choice Questions, Closed and Open Questions.
Status of prevention of postoperative delirium | Up to 2 months
  Answers of PTAiIT-members regarding measures of postoperative delirium prevention. Anonymous on-line survey including Multiple Choice Questions, Closed and Open Questions.
Status of treatment of postoperative delirium | Up to 2 months
  Answers of PTAiIT-members regarding measures of postoperative delirium treatment. Anonymous on-line survey including Multiple Choice Questions, Closed and Open Questions.

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof L Kusza, MD, PhD, Study Chair — Medical University in Poznań
Locations (2):
- Poland (2):
  - Medical University in Lublin, Lublin
  - Pomeranian Medical University, Szczecin

IPD SHARING:
Plan to Share IPD: No